CLINICAL TRIAL: NCT04401124
Title: A Descriptive Study on the Proper Management of Gastrointestinal Surgeries During the COVID-19 Pandemic, With an Emphasis on the Alteration of Surgical Protocol and Workflow
Brief Title: Status of Management of Surgery in Beijing During COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Peking University First Hospital (Other); Peking University People's Hospital (Other); Peking University Third Hospital (Other); Chinese PLA General Hospital (Other); Beijing Hospital (Other Government); Xuanwu Hospital, Beijing (Other); Peking Union Medical College Hospital (Other); Beijing Chao Yang Hospital (Other); Peking University Cancer Hospital & Institute (Other); China-Japan Friendship Hospital (Other); Peking University Shougang Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Professor, Beijing Friendship Hospital
Other Study IDs: BFH-SurgeryCovid
Record Dates: First submitted 2020-05-22; First posted 2020-05-26 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Gastric Cancer; Colorectal Cancer; Gastrointestinal Disease
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients treated at surgical emergency rooms
  Interventions: Other: no intervention
- patients receiving surgeries (both elected and emergency)
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This is a multi-centered, retrospective, observational study aimed at observing the current status of the management of gastrointestinal surgery during the COVID-19 pandemic, particularly the changes on surgery protocols and other key aspects of surgical workflow, so as to share experience with colleagues both domestic and abroad.

ELIGIBILITY:
Inclusion Criteria:

* All patients arriving at surgical emergency and all patients receiving gastrointestinal surgeries in participating centers from 2020.1.1~2020.3.31.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at surgical ER, and patients in gastrointestinal wards
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-05-25 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-06-07 (Estimated)

PRIMARY OUTCOMES:
treatment of fevers at arrival | 1 day
  proportion of patients presented with fever, proportion of patients refered to fever clinics, proportion of patients screened for COVID-19, method of screening (CT? nucleated acid test?)
treatment of post-operative fevers | 1 day
  proportion of patients on whom fever occured, proportion of patients screened for COVID-19, method of screening (CT? nucleated acid test?)
assorted surgical parameters | 1 day
  Duration of operation (≥180min/<180min); Intra-operative transfusion (Y/N); Surgical approach (Laparoscopy-involved/Open); Resection range (Non-radical/Radical); Lymph node dissection (Unknown/Not dissected/D1/D2 or above); Combined organ resection (Y/N); Post-operative complications (Y/N); Post-operative transfusion (Y/N); Post-operative hospital stay (≥7d/<7d)

SECONDARY OUTCOMES:
hospitals' protection measures and extent of implementation | 1 month
  Out-patient of surgery (Open/Closed); Emergency of surgery (Open/Closed); Fever clinic (Open/Closed); Surgical ward (Open/Closed); Functional level of surgical ward (Receive emergency surgery patients only/Receive surgery patients only/Receive all kinds of patients); Isolation ward for suspected COVID-19 patients (With/Without); Bed number in each surgical ward room (1/2/≥3); Isolation area within surgical ward (With/Without); Usage of sub-pressure operation theaters (Routinely applied/Applied for suspected patients/Never applied); Protection level of surgeons in surgical ward (No specific protection/Regular medical masks/Any of N95 mask, eye/face shields, gowns); Protection level of surgeons in ER room (No specific protection/Regular medical masks/Any of N95 mask, eye shields, face shields, gowns)

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Zhang, M.D., Principal Investigator — Beijing Friendship Hospital

IPD SHARING:
Plan to Share IPD: Undecided